CLINICAL TRIAL: NCT04787809
Title: Living Well: A Digital Acceptance and Commitment Therapy-Informed Intervention
Brief Title: Living Well: A Digital ACT Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Tyler (Other)
Responsible Party: Principal Investigator, Olga Berkout, Assistant Professor of Psychology, University of Texas at Tyler
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-FY2021-74
Record Dates: First submitted 2021-02-03; First posted 2021-03-09 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Depressive Symptoms; Anxiety; Emotional Disorders
Keywords: Acceptance and Commitment Therapy; digital mental health; depression; anxiety; emotional disorders; prevention; experiential avoidance; values
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to a treatment (digital ACT-informed intervention) or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Living Well Intervention Group (Experimental): Participants in the Living Well treatment group will receive a brief digital intervention informed by Acceptance and Commitment Therapy.
  Interventions: Behavioral: Living Well
- Control Group (No Intervention): Participants in the control group will not receive any intervention. These individuals will have the option to access the intervention at the conclusion of their study participation.

INTERVENTIONS:
Behavioral: Living Well — Living Well is a single session digital intervention that aims to decrease experiential avoidance and increase engagement in values-consistent behavior.
  Arms: Living Well Intervention Group

SUMMARY:
Depression and anxiety are frequently comorbid and share mechanisms contributing to dysfunction. Transdiagnostic approaches, such as Acceptance and Commitment Therapy, streamline intervention and allow a broader population to benefit in a cost-effective fashion. Brief ACT interventions targeting at-risk individuals have the potential to prevent negative outcomes. Delivering these in a digital format overcomes attitudinal and structural barriers to accessing treatment.

DETAILED DESCRIPTION:
Depression and anxiety disorders are among the most prevalent psychological difficulties and contribute to negative economic, social, and health outcomes. As they are frequently comorbid and share underlying mechanisms of dysfunction, many scholars have conceptualized these as a unified category of emotional disorders. Addressing processes contributing to dysfunction among individuals who are at risk for developing emotional disorders has the potential to prevent significant negative impact.

Acceptance and Commitment Therapy (ACT) has received empirical support in the treatment of depression and anxiety in a number of examinations. ACT aims to shape acceptance of challenging thoughts and feelings and engagement with areas of life one finds meaningful and important. The converse of acceptance, experiential avoidance, or the unwillingness to experience unpleasant thoughts and emotions even when doing so is maladaptive, has been predictive of symptoms of depression and anxiety. Reducing experiential avoidance and shaping alternative responses, such as acceptance and behavior consistent with one's values, termed committed action, is a promising strategy for targeting risk for emotional disorders.

Traditional means of delivering interventions fail to reach a substantial proportion of those who struggle with psychological difficulties. Barriers such as distance, time, and cost contribute to these challenges. Digital mental health interventions offer a means to overcome treatment barriers and increase access. These approaches can be delivered in individual's homes at the time of their choosing. Additionally, digital interventions can be delivered to many people at the same time, reducing cost. Support for the impact of ACT-informed digital interventions on symptoms of depression and anxiety has been obtained, suggesting that this framework is promising for reducing risk.

The goal of the current study is to compare the impact of a digital ACT-informed intervention on psychological symptoms and processes of change among individuals at risk for depression and anxiety. The following hypotheses will be evaluated:

1. Individuals in the treatment condition will experience a decrease in symptoms of depression and anxiety compared to those in the control group
2. Individuals in the treatment condition will experience a decrease in experiential avoidance and increase in values consistent behavior compared to those in the control group
3. The digital intervention will generally be rated positively
4. The relationship between cognitive fusion and treatment response will be explored

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students aged 18 or older
* Mildly to moderately elevated symptoms of depression or anxiety as reflected by DASS-21 Depression (5-10) or Anxiety scores (4-7).

Exclusion Criteria:

* Participants under the age of 18
* Severe or extremely severe scores on DASS-21 Depression (11 or greater) or Anxiety (8 or greater).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scales-21 Depression Scale repeated measure of change | pre-intervention, two week post intervention, and four week post intervention
  Depression Anxiety Stress Scales-21 (DASS-21) is a 21 item self report questionnaire assessing symptoms of depression, anxiety, and stress. The DASS-21 seven item Depression Scale will be used to assess symptoms of depression and with higher scores indicating greater depressive symptoms. Scores on the DASS-21 Depression Scale range from 0 to 21.
Depression Anxiety Stress Scales-21 Anxiety Scale repeated measure of change | pre-intervention, two week post intervention, and four week post intervention
  Depression Anxiety Stress Scales-21 (DASS-21) is a 21 item self report questionnaire assessing symptoms of depression, anxiety, and stress. The DASS-21 seven item Anxiety Scale will be used to assess symptoms of anxiety with higher scores indicating greater anxiety symptoms. Scores on the DASS-21 Anxiety Scale range from 0 to 21.
Brief Experiential Avoidance Questionnaire repeated measure of change | pre-intervention, two week post intervention, and four week post intervention
  Brief Experiential Avoidance Questionnaire (BEAQ) is a 15 item self report measure assessing experiential avoidance. Higher scores on the BEAQ indicate greater experiential avoidance. Scores on the BEAQ can range from 15 to 90.
Valuing Questionnaire-Progress Scale repeated measure of change | pre-intervention, two week post intervention, and four week post intervention
  Valuing Questionnaire-Progress Scale (VQ-P) is a five item scale assessing the extent to which one made progress towards one's values that is a part of the ten item Valuing Questionnaire. Higher scores on the VQ-P indicate greater progress towards one's values and VQ-P scores can range from 0 to 30.

OTHER OUTCOMES:
COVID-19 Impact Indicators repeated measure of change | Measured at baseline, 2 weeks post baseline, and 4 weeks post baseline
  Participants will provide information on how they have been impacted by the COVID-19 pandemic. They will respond to the question "How has the COVID-19 outbreak affected you in the past two weeks (you can select multiple options)" selecting from among 10 possible options: Diagnosed with COVID-19, worked remotely or from home more than you usually do, worked more hours than usual, worked reduced hours, was not able to work, had difficulty arranging for childcare, incurred increased costs for childcare expenses, income or pay has been reduced, not paid at all, had serious financial problems. Participants may choose between 0 and 10 possible COVID-19 impacts. These do not belong to a standardized questionnaire, but have been used by other researchers to describe the impact of COVID-19.
Cognitive Fusion Questionnaire | Measured at baseline
  The Cognitive Fusion Questionnaire is a self report measure of cognitive fusion consisting of seven items. Higher scores indicate greater cognitive fusion and scores can range from 7 to 49.
Treatment Experience/Perceived Need Questions | Measured at baseline
  Participants will respond to three questions about past experience with mental health treatment and perceived future need with yes/no responses. These questions do not belong to a standardized questionnaire, but have been used by other researchers to describe participant experience.
  In the past 12 months, did you receive therapy from a professional counselor or therapist to help you with emotional or mental health problems such as feeling sad, blue, anxious, or nervous?
  In the past 12 months, did a healthcare professional prescribe medications to help you with emotional or mental health problems such as feeling sad, blue, anxious, or nervous?
  In the past 12 months, did you think you needed help for emotional or mental health problems such as feeling sad, blue, anxious, or nervous?

CONTACTS AND LOCATIONS:
Overall Officials: Olga Berkout, PhD, Principal Investigator — University of Texas at Tyler
Locations (1):
- UT Tyler, Tyler, Texas, United States

IPD SHARING:
Plan to Share IPD: No